CLINICAL TRIAL: NCT02122094
Title: Implementation of a Sexual Health Intervention for YMSM in Two Vietnamese Cities
Brief Title: Implementation of a Sexual Health Intervention for Young Men Who Have Sex With Men (MSM) in Two Vietnamese Cities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Hanoi Medical University (Other); University of Puerto Rico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01DA033673 (NIH)
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2015-10

CONDITIONS: HIV; Chlamydia; Gonorrhea; Syphilis; Hepatitis C
MeSH Terms: conditions — Chlamydia Infections; Gonorrhea; Syphilis; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sexual Health Promotion Intervention (Experimental): The SHP Intervention consists of seven core and five optional modules covering topics related to sexual health. It is delivered in both community (outreach) settings and i clinic-based settings.
  Interventions: Behavioral: Sexual Health Promotion Intervention

INTERVENTIONS:
Behavioral: Sexual Health Promotion Intervention — The seven core modules are 1) the Importance of Sexual Health, 2) Sexual Diversity, 3) HIV and other STIs, 4) Behavioral Risk and Risk Reduction, 5) Alcohol and Drugs, 6) Stigma and 7) Health Seeking Practices. The five optional modules are 1) HIV Treatment and Adherence, 2) Stress Reduction, 3) HIV Status Disclosure, 4) MSM/Gay Disclosure, and 5) Other Sexual Health Concerns

SUMMARY:
This study seeks to implement a sexual health promotion intervention for male sex workers in Hanoi and Ho Chi Minh City, Vietnam. The study hypothesis is that this intervention will increase testing, treatment and vaccination for sexually transmitted infections, including intentions of participants to engage in these services beyond the conclusion of the intervention. At the community level, the study hypothesis is that male sex workers will be more aware of sexual health care and more likely to access these services in the future.

DETAILED DESCRIPTION:
The intervention is administered in community and clinic settings. The full intervention consists of seven core modules: Sexual Health, Sexual Diversity, HIV/STI Transmission, Behavioral Risk and Risk Reduction, Alcohol and Drugs, Stigma, and HIV/STI and Health Seeking Practices. In the community, outreach is conducted by Health Educators to deliver the intervention modules that young men express and interest in, as well as to provide risk reduction materials including condoms and lubricant. Study interviewers conduct a cross-sectional interview of young male sex workers in community venues (the interviewers and health educators are never present in a venue at the same time), and a random sample of interviewees are invited to a local clinic, where they receive a more detailed interview, the full intervention (delivered one on one by a Health Educator and including all seven modules), a clinical exam, testing for HIV and other STIs (HBV, HCV, gonorrhea, syphilis, chlamydia), onsite treatment, vaccination and referral, and a post-intevention assessment.

ELIGIBILITY:
Inclusion Criteria:

* Born biologically male; age 16-29; exchanged sex for money or other material goods with another man in the past 90 days

Exclusion Criteria:

* inability to provide informed consent

Ages: 16 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1166 (Actual)
Dates: Start 2013-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Acceptance of testing | 2 hours
  Participants in the clinic-based Sexual Health Promotion intervention will accept offer of testing for chlamydia, gonorrhea, syphilis, HIV, HBV and Hepatitis C Virus.
Return for test results | two weeks
  Participants in the clinic-based Sexual Health Promotion intervention will return for their test results
Intention to access health services | two years
  Participants who receive the community-based Sexual Health Promotion intervention will report intent to access health services for Sexually Transmitted Infection testing, treatment and vaccination

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Hanoi Medical University, Hanoi, Hanoi
  - Center for Applied Research on Men and Health (CARMAH), Ho Chi Minh City, Ho Chi Minh CIty